CLINICAL TRIAL: NCT06316674
Title: The Malleability of Body Representation in Anorexia Nervosa: the Sixth Finger Illusion
Acronym: SESTODITO_AN
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Heriot-Watt University (Other); Birkbeck, University of London (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: 03C304
Record Dates: First submitted 2024-02-28; First posted 2024-03-18 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa (AN): People affected by AN (DSM5); female, age 18-55, BMI ≤ 17.5 Kg/m2
  Interventions: Behavioral: sixth finger illusion
- Healthy controls (HC): female, age 18-55, BMI between 18.5 Kg/m2 and 25 Kg/m2
  Interventions: Behavioral: sixth finger illusion

INTERVENTIONS:
Behavioral: sixth finger illusion — Participants will undertake the sixth finger illusion that is a body illusion which elicits the presence of an extra numerary finger due to visuo-tactile stimulation.

SUMMARY:
Body representation can be explored using behavioural tasks such as motor imagery tasks as well as body illusions.

In both cases, evidence from studies on healthy individuals as well as patients with lesions to the central nervous system show that body representation is not set in stone: how we imagine our bodies is a dynamic and continuously updated process, to reflect changes in our own body as well as the environment.

In anorexia nervosa the representation of the body is very different from that of healthy individuals: the representation is more malleable, and easier to manipulate, while at the same time being more detached from physical constraints. These features of body representation in anorexia nervosa might contribute to the persistence of symptoms and to relapses too. Body representation has clear implications for treatment of anorexia nervosa too.

The study aims at evaluating the presence of differences in the malleability of the body representation, explored through the illusion of the sixth finger, between a group of people with AN and a group of normal weight people, taking into account the biomechanical constraints that characterize the physical and mentally represented body.

DETAILED DESCRIPTION:
The ability to imagine our body in our mind is called body representation. This ability is grounded in sensory and perceptual process and it is crucial to plan action, to interact with the environment and so on. Body representation can be explored using behavioural tasks such as motor imagery tasks as well as body illusions.

Evidence from healthy individuals shows that we depend on physical constraints when we imagine actions we can do with our body: we are faster and more accurate in imagining an action that we can really perform. This phenomenon is called "biomechanical constraints effect" and it is an index that our brain is performing motor imagery. When a lesion occurs to the spinal cord, for example, this effect is not present anymore, supporting the idea that what occurs in our brain is strongly dependent on what we can do in the real word. This dependency from the real word, however, does not mean that the representation of the body in the mind is an exact copy of the physical body. For example, findings from experiments using body illusions show that we have a distorted representation of our body, even in absence of any lesion. Overall, evidence from body illusions in healthy individuals shows that we tend to overestimate features when we imagine our body, width in particular compared to length and height.

In both cases, evidence from studies on healthy individuals as well as patients with lesions to the central nervous system show that body representation is not set in stone: how we imagine our bodies is a dynamic and continuously updated process, to reflect changes in our own body as well as the environment.

Recent studies suggest that body representation is quite different in conditions that affect the body even in absence of central nervous system or brain impairments, such as anorexia nervosa. In patients affected by anorexia nervosa, motor imagery does not occur, and patients treat their body like it is an object. Similarly, when subjected to illusions of ownership, patients with anorexia nervosa experience the illusion more strongly than healthy individuals.

In anorexia nervosa the representation of the body is very different from that of healthy individuals: the representation is more malleable, and easier to manipulate, while at the same time being more detached from physical constraints. These features of body representation in anorexia nervosa might contribute to the persistence of symptoms and to relapses too. Body representation has clear implications for treatment of anorexia nervosa too.

The study aims at evaluating the presence of differences in the malleability of the body representation, explored through the illusion of the sixth finger, between a group of people with AN and a group of normal weight people, taking into account the biomechanical constraints that characterize the physical and mentally represented body.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-55 years
* bmi ≤ 17.5 Kg/m2 for AN and BMI between 18.5 Kg/m2 e 25 Kg/m2 for healthy controls

Exclusion Criteria:

* psychopathologies related to psychosis or brain injury lesions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female Anorexia Nervosa patients and female healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Sixth finger illusion questionnaire | Through study completion, an average of 1 year
  Participants are asked to answer to a 6 questions questionnaire based on a likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico italiano IRCSS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brusa F, Kretzschmar L, Magnani FG, Turner G, Garraffa M, Sedda A. Talking with hands: body representation in British Sign Language users. Exp Brain Res. 2021 Mar;239(3):731-744. doi: 10.1007/s00221-020-06013-4. Epub 2021 Jan 3. PMID 33392694
- [Background] Brusa F, Suphi Erden M, Sedda A. Exploring the role of disgust in hands and feet laterality judgement tasks. Q J Exp Psychol (Hove). 2024 Jul;77(7):1418-1429. doi: 10.1177/17470218231207336. Epub 2023 Nov 3. PMID 37800303
- [Background] de Vignemont F. Body schema and body image--pros and cons. Neuropsychologia. 2010 Feb;48(3):669-80. doi: 10.1016/j.neuropsychologia.2009.09.022. Epub 2009 Sep 26. PMID 19786038
- [Background] Eshkevari E, Rieger E, Longo MR, Haggard P, Treasure J. Increased plasticity of the bodily self in eating disorders. Psychol Med. 2012 Apr;42(4):819-28. doi: 10.1017/S0033291711002091. Epub 2011 Oct 5. PMID 22017964
- [Background] Eshkevari E, Rieger E, Longo MR, Haggard P, Treasure J. Persistent body image disturbance following recovery from eating disorders. Int J Eat Disord. 2014 May;47(4):400-9. doi: 10.1002/eat.22219. Epub 2013 Nov 18. PMID 24243423
- [Background] Fiori F, Sedda A, Ferre ER, Toraldo A, Querzola M, Pasotti F, Ovadia D, Piroddi C, Dell'Aquila R, Redaelli T, Bottini G. Motor imagery in spinal cord injury patients: moving makes the difference. J Neuropsychol. 2014 Sep;8(2):199-215. doi: 10.1111/jnp.12020. Epub 2013 May 15. PMID 23672438
- [Background] Holmes NP, Spence C. The body schema and the multisensory representation(s) of peripersonal space. Cogn Process. 2004 Jun;5(2):94-105. doi: 10.1007/s10339-004-0013-3. PMID 16467906
- [Background] Scarpina F, Bastoni I, Villa V, Mendolicchio L, Castelnuovo G, Mauro L, Sedda A. Self-perception in anorexia nervosa: When the body becomes an object. Neuropsychologia. 2022 Feb 10;166:108158. doi: 10.1016/j.neuropsychologia.2022.108158. Epub 2022 Jan 14. PMID 35033502